CLINICAL TRIAL: NCT00679003
Title: Psychosocial Intervention for Children With IBD
Brief Title: Managing Inflammatory Bowel Disease
Acronym: Managing IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Seattle Children's Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rona Levy, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRMC12395; 1R01HD050345-01A2 (NIH)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease; Ulcerative colitis; Inflammatory bowel disease; Illness behavior; Cognitive behavioral therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Illness Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Social learning and cognitive behavioral therapy (SLCBT)
  Interventions: Behavioral: SLCBT
- 2 (Active Comparator): Education and support (ES)
  Interventions: Behavioral: ES

INTERVENTIONS:
Behavioral: SLCBT — Social learning and cognitive behavioral therapy
  Arms: 1
Behavioral: ES — Education and support (information about nutrition and gastrointestinal system)
  Arms: 2

SUMMARY:
Inflammatory Bowel Disease (Crohn's disease and ulcerative colitis) often results in significant life disruption, hospitalization and surgery. While psychosocial factors are not believed to cause IBD, such factors can contribute to the ability of individuals with IBD to cope with the disease, and ineffective coping may lead to the exacerbation of IBD symptoms. The goal of this study is to evaluate the efficacy of a social learning and cognitive behavior therapy approach for treating children with IBD. The primary outcomes of interest are IBD symptoms, medical visits, quality of life, and overall disability.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (Crohn's and ulcerative colitis; IBD), a serious medical condition that affects children and adolescents, is often associated with high rates of health care utilization and disability, including school absences. While psychosocial factors are not believed to cause IBD, research suggests that they may increase illness-related dysfunction. Prior studies suggest that response to chronic illness is, in part, acquired during childhood through social learning processes and may be modified with psychosocial interventions. This randomized controlled trial will compare a social learning and cognitive behavior therapy (SLCBT) treatment to an education and support condition (ES). 180 children with IBD will be recruited and followed for 12 months. It is hypothesized that SLCBT participants, compared to those in the ES condition, will, at one-year follow-up: 1) exhibit greater decreases in IBD symptoms, medical visits for IBD, and functional disability, and greater increases in quality of life; 2) demonstrate greater use of cognitive coping, relaxation and stress management skills, and their parents will demonstrate greater reductions in maladaptive responses to illness behavior; and 3) exhibit greater reductions in anxiety, depression, and somatization. Results will lead to innovative interventions for IBD and other chronic childhood medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Child has been diagnosed for at least 3 months
* Child age is 8-17
* Child has lived with primary caregiver full-time for at least the past 5 years and for at least half of his/ her lifetime
* Child is medically approved to engage in normal daily activities

Exclusion Criteria:

* Chronic disease other than IBD (e.g., pancreatitis, diabetes, epilepsy)
* Major surgery in past year unrelated to IBD
* Developmental disabilities that require full-time special education or that impair ability to respond to treatment

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2007-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Functional Disability Inventory | Baseline (1 week pre-treatment), 1 week post-treatment, 3 months, 6 months and 12-months post-treatment

SECONDARY OUTCOMES:
School absences | Baseline, 3 months, 6 months and 12 months post-treatment
Health care utilization for IBD | Baseline, 3 months, 6 months and 12 months post-treatment
Pediatric Quality of Life | Baseline (1 week pre-treatment), 1 week post-treatment, 3 months, 6 months and 12 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rona L Levy, MSW, PhD, MPH, Principal Investigator — University of Washington; Tasha B Murphy, PhD, Study Director — University of Washington

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] van Tilburg MAL, Claar RL, Romano JM, Langer SL, Drossman DA, Whitehead WE, Abdullah B, Levy RL. Psychological Factors May Play an Important Role in Pediatric Crohn's Disease Symptoms and Disability. J Pediatr. 2017 May;184:94-100.e1. doi: 10.1016/j.jpeds.2017.01.058. Epub 2017 Feb 24. PMID 28238483